CLINICAL TRIAL: NCT00277108
Title: Open Label Variable Dose Escitalopram (Lexapro) in the Treatment of Patients With Postpartum Major Depression: A Pilot Study
Brief Title: Lexapro in the Treatment of Patients With Postpartum Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Forest Laboratories (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LXP-MD80
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2008-11-06 (Estimated); Status verified 2008-11

CONDITIONS: Postpartum Depression
Keywords: postpartum depression; postnatal depression; PPD
MeSH Terms: conditions — Depression, Postpartum | interventions — Escitalopram

INTERVENTIONS:
Drug: Escitalopram (Lexapro)

SUMMARY:
The purpose of this study is to determine if Escitalopram (Lexapro) is effective in the treatment of postpartum depression.

DETAILED DESCRIPTION:
Primary objectives: Remission of Major Depression: To determine the efficacy of a flexibly titrated dose of Escitalopram (10mg to 20 mg) in the treatment of women with postpartum depression. The primary outcome measure will be remission of major depression, defined as a score of 12 or less on the Montgomery-Asberg Depression Scale. A score of 7 or less on the Hamilton Depression Scale (21 item) will be used as a secondary measure of remission. The null hypothesis is that flexibly dosed Escitalopram does not lead to remission of major depression based on total MADRS scores after 8 weeks of treatment.

Secondary objectives:

1. To determine if treatment with Escitalopram is effective in achieving significant reduction in symptoms of postpartum depression as measured on several instruments: HAM-D 21, CGI, Beck Depression Inventory, Edinburgh Postnatal Depression Scale. Specifically, a response will be defined as a reduction of the total scores of 50% or more from baseline on the MADRS or HAM-D 21.
2. To determine the tolerability, safety and some dosing considerations for Escitalopram in this special subpopulation of depressed patients. Adverse events data (clinical and laboratory), compliance and early termination will be used as outcome measures.
3. To determine in a post-hoc analysis if pre-study anxiety levels as measured with HAM-A correlate with primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Biological mothers of infants ages 2 weeks to 12 months of age
2. Age 18 and over
3. Must understand and speak English well enough to read and provide written informed consent, complete written questionnaires and complete the SCID.
4. The primary Axis I diagnosis, as determined by the SCID, must meet the DSM-IV criteria for Unipolar Major Depression, Single or Recurrent, Moderate to Severe. Onset of depression must occur within pregnancy to the first 12 months following childbirth. Concurrent diagnoses of anxiety disorders including obsessive compulsive disorder, panic disorder, specific phobias, generalized anxiety disorder, and post-traumatic stress disorder will be allowed if they are not the primary diagnosis.
5. The subject must receive a MADRS total score of > 22 at screening and at the baseline visit and a total score of >17 on the HAM-D at the baseline visit.
6. The subject must be able to comply with instructions and be capable of participating in an 8 week study.

   -

Exclusion Criteria:

1. Under 18 years of age.
2. Subjects who are breastfeeding.
3. History of Bipolar Disorder, Schizoaffective Disorder, Schizophrenia.
4. History of any DSM-IV Axis II diagnosis, which in the investigator's opinion, would interfere with compliance of the protocol.
5. History of alcohol or drug abuse or dependence in the last year.
6. Treatment with other psychotropic drugs except permissible concomitants.
7. Current severe psychiatric symptoms requiring psychiatric hospitalization, current psychosis or suicidal, homicidal potential.
8. History of intolerance to or hypersensitivity to Citalopram.
9. Subjects whose depressions are known to be unresponsive to Escitalopram.
10. Subjects who are pregnant or who intend to become pregnant during the course of the study.
11. Subjects who have any medical or neurological disorder that in the investigators' opinion may contribute to depression.
12. Subjects who have started psychotherapy within three months prior to baseline or who intend to start psychotherapy during the study.

    -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2004-02; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be remission of major depression, defined as a score of 12 or less on the Montgomery-Asberg Depression Scale.

SECONDARY OUTCOMES:
A score of 7 or less on the Hamilton Depression Scale (21 item) will be used as a secondary measure of remission.

CONTACTS AND LOCATIONS:
Overall Officials: Linda H Chaudron, MD, MS, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States